CLINICAL TRIAL: NCT03091608
Title: A Registry Study to Surveil Early Liver Injuries Caused by Xianlin Gubao Granule (XLGB Granule)
Brief Title: Surveillance for Early Liver Injuries Caused by Xianlin Gubao Granule
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Principal Investigator, Xiaohe Xiao, Director, Beijing 302 Hospital
Other Study IDs: 302-xxh-XLGBG
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Drug-Induced Liver Injury
Keywords: Drug-Induced Liver Injury
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Biospecimen Retention: Samples With DNA — serum, plasma, histology and urine.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The individuals taking XLGB Granule: The overall individuals taking XLGB Granule with recommended dosage and achieving the inclusion criteria.

SUMMARY:
This is a prospective registry study to surveil early liver injuries caused by Xianlin Gubao Granule (XLGB Granule) through a non-intervention observational way. And attempt to establish a predictive model to screen susceptibilities to XLGB Granule.

DETAILED DESCRIPTION:
The primary objectives of this study include:

(i) The detection of patients with serum liver biochemistry abnormalities within 8 weeks after intake of XLGB Granule; (ii) The record of overall individuals with demographics, underlying diseases, physical status, medication information, clinical laboratory index, and so on; (iii) The specimen collection of surveiled individuals. (iv) The attempt to establish a predictive model to screen susceptibilities to XLGB Granule.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals in accordance with indications for XLGB Granule, including osteoporosis, fracture, osteoarthritis, aseptic necrosis of bone and climacteric;
2. The age range of 18 to 70 years;
3. Individuals taking XLGB Granule over 2 weeks;
4. Abnormalities of serum liver biochemistry achieving one of the criteria as follows:

   (i) alanine aminotransaminase (ALT) or aspartate transaminase (AST) ≥2 folds of upper limit of normal (ULN); (ii) total bilirubin (TBiL) ≥ 2 ULN; (iii) alkaline phosphatase (ALP) ≥ 2 ULN;
5. Individuals can provide informed consent form.

Exclusion Criteria:

1. Individuals without indications for XLGB Granule;
2. Unconformity to the XLGB Granule drug label;
3. Individual taking XLGB Granule less than 2 weeks;
4. Individuals taking other hepatotoxic drugs combined with XLGB Granule, simultaneously;
5. Unconformity to the diagnostic standard for herb-induced liver injury (the Guideline for Diagnosis and Treatment of Herb-induced Liver Injury, RPGIP-2016CN003）.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample and primary care clinic.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-03-25 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
The detection of patients with serum liver biochemistry abnormalities within 8 weeks after intake of XLGB Granule. | participants will be followed duration intake of XLGB Granule, an expected average within 8 weeks
  The detection of patients with serum liver biochemistry abnormalities within 8 weeks after intake of XLGB Granule.

SECONDARY OUTCOMES:
Clinical features of early liver injuries caused by XLGB Granule assessed by serum parameters of liver function. | participants will be followed duration intake of XLGB Granule, an expected average of 8 weeks
  Clinical features of early liver injuries caused by XLGB Granule assessed by serum parameters of liver function.

OTHER OUTCOMES:
Disease progression of early liver injuries caused by XLGB Granule, i.e. death, liver failure, chronic DILI, recovery. | 8 weeks
  Disease progression of early liver injuries caused by XLGB Granule, i.e. death, liver failure, chronic DILI, recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-he Xiao, Study Director — 302 Military Hospital
Locations (1):
- 302 Military Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided